CLINICAL TRIAL: NCT03678623
Title: Exploring the Impact of Standing on the Musculoskeletal System of Sedentary-workers
Brief Title: The Impact of Prolonged Standing on Musculoskeletal Pain
Status: Completed | Type: Observational
Sponsor: Universidade da Coruña (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Beatriz Rodríguez-Romero, Principal Investigator. PhD, MSc, PT. Lecturer at Faculty of Physiotherapy, Universidade da Coruña., Universidade da Coruña
Other Study IDs: Standing-musculoskeletal pain
Record Dates: First submitted 2018-09-09; First posted 2018-09-19 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Musculoskeletal Pain; Occupational Exposure; Office Workers
Keywords: Musculoskeletal Pain; Occupational Exposure; Predictive value of tests; Back muscles
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Office-based workers: Individuals working in an office environment with their main tasks involving use of a computer, reading, phoning, making presentations and participating in meetings, who perform more than 30 hours per week mostly sitting at a computer.

SUMMARY:
This is a cross-sectional and prospective cohort study using a biopsychosocial approach to investigate office workers at risk of standing-induced musculoskeletal pain. The purpose of this study is to determine which factors are associated with developing or worsening of musculoskeletal pain (changes in the Visual Analogue Scale from baseline) during a 60 minute standing paradigm.

DETAILED DESCRIPTION:
Background/rationale

There is growing national and international evidence for the negative health impact of sedentary behaviour at work. A strategy being increasingly adopted to reduce prolonged sitting is to spend some of the work day in standing. However, for some adults, prolonged standing is associated with the development of musculoskeletal pain. We are investigating which factors are associated with developing of musculoskeletal pain during standing when using a height-adjustable desk. Previous studies have used an induced-pain paradigm to understand risk factors for developing musculoskeletal pain during a prolonged standing task that simulates the work environment (standing paradigm). Identifying those office workers who are at risk of developing musculoskeletal pain during standing will provide information to guide health professionals and individuals in making decisions about optimal workstation design.

Objectives and hypothesis

* Cross-sectional study: Identify which factors are associated (demographic, physical, psychological and work-related factors) with standing-induced musculoskeletal pain in office workers during a standing paradigm.
* Prospective cohort study: Identify incidence/prevalence and risk factors of low back pain, and disability associated with low back pain in office workers in a 1-year prospective cohort.

Methods

* Setting, locations and relevant dates: testing is conducted in the University of Queensland (Brisbane, Australia). Data collection commenced in May of 2018 until 30th of April of 2019 (cross-sectional study); and follow-up is from June of 2018 until 30th of April of 2020 (prospective cohort study).
* Participants: recruitment is through posting flyers on campus of The University of Queensland; through the weekly electronic university staff newsletter at this University; and through Facebook announcements. Interested participants were directed to an online questionnaire (hosted by Survey Monkey) to determine eligibility. Participants meeting the eligibility criteria were contacted via email to schedule an appointment.
* Variables: see "outcomes measures".
* Study size: a convenience sample of 40 office workers will be recruited. Based on previous studies that have compared developers and non-developers of standing-induced low back pain, this sample size was considered sufficient to detect a significant difference in some of the physical outcome measures such as lumbar lordosis (Sorensen et al. 2015a); trunk muscle activation (Ringheim et al. 2015) and active hip abduction (Nelson-Wong et al. 2008).
* Statistical analysis: subjects will be separated into Pain Developers (PDs) and Non-Pain Developers (NPDs). A Chi-square analysis or a Fisher's Exact test will be conducted to test for differences in the distribution of qualitative and proportional variables in PDs and NPDs. Independent groups t-tests, will be conducted to test for differences in quantitative variables between PDs and NPDs. A Pearson correlation coefficient and one-way analysis of variance test will be conducted to test for differences for average Visual Analogue Score (VAS). A simple linear regression analysis will be performed to examine the degree to which biopsychosocial variables predict PDs. Statistical analyses will be performed in SPSS version 24 (IBM, Armonk, NY).Statistical significance for all tests will be set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Office-based workers who perform more than 30 hours per week mostly sitting at a computer,
* With aged 18 or above.

Exclusion Criteria:

* not office-based workers,
* pregnant or less than six months postpartum,
* had experienced any major trauma or had surgery to the spine or lower limb over the last 12 months,
* had been diagnosed with any neurological or systematic pathology (such as rheumatoid arthritis, multiple sclerosis or ankyloses spondylitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Office-based workers, defined as individuals working in an office environment with their main tasks involving use of a computer, reading, phoning, making presentations and participating in meetings, who perform more than 30 hours per week mostly sitting at a computer.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Standing Tolerance Test (STT) | Baseline
  The Standing Tolerance Test consists of participants standing for 1-hour while performing computer tasks using a workstation table.They are required to stand in a confined working area marked on the ground (60x122 cm). During the 1-h period, participants are instructed to adopt a comfortable position that they would normally use if they are to stand for a prolonged period of time. The participant are not allowed to lean on the workstation in any way. The working surface for each participant is adjusted to a height of 5 cm below elbow height. Participants rate their musculoskeletal symptoms intensity on a scale from 0 to 100 mm visual analogue scale (VAS) prior to the start of, every 15 minutes during, and at the end of the 1-h standing period. Based on their VAS rating for spine, lower and upper limb, they are classified either as a Pain Developers (PDs) if they report a change in VAS of 1 or more from baseline on 0-100 scale (whatever baseline is) or a Non-Pain Developers (NPDs).

SECONDARY OUTCOMES:
Demographic characteristics: | Baseline
  Date of birth, gender, height, weight and smoking habits are recorded
Occupational characteristics: Occupational Sitting and Physical Activity Questionnaire (OSPAQ) | Baseline
  Questions are about the time spent on activities at work over the past seven days, involving sitting, standing, walking and physically demanding tasks.
  1. How many hours did you work in the last 7 days? _____ Hours
  2. During the last 7 days, how many days were you at work? _____ Days
  3. How would you describe your typical work day in the last 7 days? (This involves only your work day, and does not include travel to and from work, or what you did in your leisure time) Please ensure your answers add up to 100.
     1. Sitting :____%
     2. Standing:____%
     3. Walking: ____%
     4. Heavy Labour or physically demanding tasks: ____% Total:____% (100%)
  Scoring:
  Minutes sitting at work per week = Item 1 * Item 3a Minutes sitting per workday = (Item 1/Item 2) * Item 3a Similar calculations can be done for standing, walking, and heavy labour.
Occupational characteristics: questions about using sit-stand workstation | Baseline
  i) Do you usually use a sit-stand workstation? Yes/No ii) How long (in month) have you had one? iii) What percentage of day do you use your sit-stand workstation?
Occupational characteristics: Abbreviated Job Content Questionnaire (JCQ) & Job Satisfaction | Baseline
  JCQ comprises 18 items measuring 5 dimensions related with psychosocial job characteristics: decision latitude, decision authority, psychological job demands, social support and physical job demands.
  Range of scores:
  * Skill discretion: 12-48
  * Decision authority: 12-48
  * Phychological job demands: 3-12
  * Social Support: 4-16
  * Physical demands: 2-8 *Job control = skill discretion + decision authority: 24-96
  Dichotomised physical demand and job control are combined to create four categories:
  * low strain: low demand and high control
  * active job: high demand and high control
  * passive job: low demand and low control
  * job strain: high demand and low control
  Job Satisfaction: comprises 1 question:
  "How satisfied are you with your work in general"?
  1. extremely dissatisfied
  2. very dissatisfied
  3. rather dissatisfied
  4. more or less satisfied
  5. rather satisfied
  6. very satisfied
  7. extremely satisfied
International Physical Activity Questionnaire (IPAQ)-Short Form | Baseline
  Questions are about physical activities(PA) (vigorous, moderate, walking) that people do as part of their everyday lives; and about the time they spent being physically active in the last 7-days. Values are computed for walking(W), moderate-intensity-activities(M), vigorous-intensity-activities(V) and a combined total physical activity score. Scores are expressed in MET-minutes/week (METs). The following values are used for the analysis: W=3.3 METs; M=4.0 METs; V=8.0 METs. There are 3 levels of PA proposed to classify populations: Low: individuals who not meet criteria for categories 2 or 3. Moderate: a)3 or more days of V of at least 20 min per day; b)5 or more days of M and/or W of at least 30-min per day; c)5 or more days of any combination of W, M or V achieving a minimum total PA of at least 600-METs. High: a)V on at least 3 days achieving a minimum total PA of at least 1500-METs; b)7 or more days of any combination of W, M or V achieving a minimum total PA of at least 3000-METs.
Quality of life related to health: SF12 questionnaire | Baseline
  SF12 questionnaire. This questionnaire ask about the generic health status in 8 domains: physical function, role physical, body pain, general health, vitality, social function, role emotional and mental health. It is a shorter version of SF-36.
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Both Physical and Mental Health Composite Scales combine the 12 items in such a way that they compare to a national norm with a mean score of 50.0 and a standard deviation of 10.0.
  A positive score means the person is healthier than average. A negative score means a person is less healthy than average.
Prevalence of musculoskeletal pain: Nordic Musculoskeletal Questionnaire (NMQ) | Baseline
  An abbreviated version of NMQ is used, which consists of a rear view of the human body, divided into 9 anatomical regions (3 each on the upper limbs, spine and lower limbs), asking about presence of musculoskeletal pain during the last year, the last month and today.
  All response options are dichotomous (yes/no). Questions are ordered in such a way that those relating to the respondents' last year are asked first, followed by prevalence questions about last month and today. Key words are highlighted in bold. Respondents are asked to answer all questions for a body region before progressing to the next region (ie, horizontally rather than vertically). If the respondent answer no for question relating to annual prevalence, they are directed to go on to the next body region and all remaining questions for that region are automatically coded as negative responses.
Symptom intensity level of musculoskeletal pain: Visual Analogue Scale (VAS) | Baseline
  The musculoskeletal intensity in 9 regions, over the previous 7 days, is measured with the VAS.
  VAS is a continuous scale comprised of a horizontal line, 10 centimetres (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst imaginable pain" (score of 100-mm scale).
Disability due to low back pain: | Baseline
  Oswestry Disability Questionnaire. Lumbar functional disability is measured using this outcome assessment. It contains 10 questions about: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and traveling. The total score is expressed as a percentage (from 0 to 100). Between 0% and 20% is interpreted as minimal disability; 21% to 40% as moderate disability; 41% to 60% as severe disability; 61% to 80% as crippled; and from 81% to 100% as bed-bound, or exaggerating their symptoms.
Catastrophizing thoughts related with pain | Baseline
  Pain Catastrophizing Scale (PCS). This scale consists of 13 statements describing different thoughts and feelings that may be associated with pain. The participant indicate the degree to which they have these thoughts and feeling is it a 5 point scale from "not at all" to "all the time" about the experiences with painful situations.
Thoracic and lumbar curve | Baseline
  The flexible ruler, length 60 cm is placed over the spinous processes of the thoracic and lumbar spine so that it follows the contour of the spinal curves, from C7 to the posterior superior iliac spine (PSIS). Spinal processes of the C7 and T12 vertebras, and PSIS are identified and marked. The flexicurve is marked at C7, T12 and S2 level; then it is carefully removed, placed on a stable surface, and the internal edge (the side of the flexicurve in contact with the skin) is traced onto graph paper. Two measurements are obtained from the flexicurve.
Motor Control Impairment test: Active hip abduction test | Baseline
  a) Active Hip Abduction test: Side-lying position. Participants are instructed to raise their top leg towards the ceiling as far as they can. The side to be tested first is randomized. Examiner score as: 0 = Able to maintain position; 1 = Minimal loss; 2 = Moderate loss; 3 = Severe loss of pelvis position in the frontal plane.
Motor Control Impairment test: Active straight leg raise test | Baseline
  b) Active Straight Leg Raise test (ASLR test): Supine position, with straight legs and feet 20 cm apart. Subject is instructed to raise a straight leg 20 cm above the table. Scoring on a 6-point scale (range 0-5). Scores of both sides are added.
Motor Control Impairment test: Prone knee flexion test | Baseline
  c) Prone Knee Flexion test: Prone position. Instruction is "bend your knee as far as you can without moving your back". Scoring: a) correct: active knee flexion at least 90° without movement of the low back and pelvis; b) incorrect: by the knee flexion low back does not stay neutral maintained but moves in extension or rotation.
Endurance tests of the trunk muscles (McGill's protocol): Sorensen test | Baseline
  Trunk endurance test (McGill´s protocol 1999):
  a) Sorensen test: The patient lies on the examining table in the prone position with the upper edge of the iliac crests aligned with the edge of the table. The lower body is fixed to the table by three straps, located around the pelvis, knees, and ankles, respectively.
  With the arms folded across the chest, the patient is asked to isometrically maintain the upper body in a horizontal position. The time during which the patient keeps the upper body straight and horizontal is recorded. In patients who experience no difficulty in holding the position, the test is stopped after 240 s.
Endurance tests of the trunk muscles (McGill's protocol): Abdominal endurance test | Baseline
  Trunk endurance test (McGill´s protocol 1999):
  b) Abdominal endurance test: This test is performed by having the subject sit on a test bench. Both the knees and hips are flexed at 90° and the feet are fixed to the bench with a strap. The arms crossed over the chest. At the position of 60° trunk flexion, the support of the trunk is then removed and the participant hold the position for as long as possible. The test is terminated when the participant is no longer able to hold the position.
Endurance tests of the trunk muscles (McGill's protocol): Side bridge test | Baseline
  Trunk endurance test (McGill´s protocol 1999):
  c) Side bridge test: The side bridge test (right and left side) are performed in the side-lying position on a mat. The participant's knees are extended with the top foot placed in front of the lower foot. The participant supports their weight only on their lower elbow and feet while lifting their hips off the mat. The test is stopped when the side-lying position is lost or when the hips returned to the mat.
Endurance tests of the trunk and hip muscles: Supine Bridge Test | Baseline
  Supine Bridge Test:
  subject is on the examination table in the supine position, with knees flexed 90 degrees and the soles of the feet on the floor.The hands are positioned by the ears. Subjects are instructed to raise the pelvis from the floor so that the shoulders, hips, and knees are maintained in a straight line. The time is held and timed until the position can no longer be maintained.
Endurance tests of the hip muscles: Abductor Hip Endurance Test | Baseline
  Abductor Hip Endurance Test:
  in the side-lying position with the evaluated hip placed superiorly in neutral alignment and with the pelvis stabilized by straps. External weight of 7.5% of body mass, is placed on the ankle of the evaluated limb. A inclinometer is strapped 10 cm superior to the lateral femoral condyle. The subject is instructed to isometrically hold the limb in a horizontal position. The time is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Venerina Johnston, PhD, Study Chair — The University of Queensland
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neuhaus M, Eakin EG, Straker L, Owen N, Dunstan DW, Reid N, Healy GN. Reducing occupational sedentary time: a systematic review and meta-analysis of evidence on activity-permissive workstations. Obes Rev. 2014 Oct;15(10):822-38. doi: 10.1111/obr.12201. Epub 2014 Jul 11. PMID 25040784
- [Background] Coenen P, Parry S, Willenberg L, Shi JW, Romero L, Blackwood DM, Healy GN, Dunstan DW, Straker LM. Associations of prolonged standing with musculoskeletal symptoms-A systematic review of laboratory studies. Gait Posture. 2017 Oct;58:310-318. doi: 10.1016/j.gaitpost.2017.08.024. Epub 2017 Aug 24. PMID 28863296
- [Background] Sorensen CJ, Johnson MB, Callaghan JP, George SZ, Van Dillen LR. Validity of a Paradigm for Low Back Pain Symptom Development During Prolonged Standing. Clin J Pain. 2015 Jul;31(7):652-9. doi: 10.1097/AJP.0000000000000148. PMID 25171636
- [Background] Marshall PW, Patel H, Callaghan JP. Gluteus medius strength, endurance, and co-activation in the development of low back pain during prolonged standing. Hum Mov Sci. 2011 Feb;30(1):63-73. doi: 10.1016/j.humov.2010.08.017. Epub 2011 Jan 11. PMID 21227522
- [Background] Nelson-Wong E, Gregory DE, Winter DA, Callaghan JP. Gluteus medius muscle activation patterns as a predictor of low back pain during standing. Clin Biomech (Bristol). 2008 Jun;23(5):545-53. doi: 10.1016/j.clinbiomech.2008.01.002. Epub 2008 Feb 20. PMID 18282648
- [Background] Zamkova MA, Krivitskaia EI. [The effect of radiation by erythema-uviol lamps on the working capacity of students]. Gig Sanit. 1966 Apr;31(4):41-4. No abstract available. Russian. PMID 4384659
- [Background] Sorensen CJ, Norton BJ, Callaghan JP, Hwang CT, Van Dillen LR. Is lumbar lordosis related to low back pain development during prolonged standing? Man Ther. 2015 Aug;20(4):553-7. doi: 10.1016/j.math.2015.01.001. Epub 2015 Jan 14. PMID 25637464
- [Background] Ringheim I, Austein H, Indahl A, Roeleveld K. Postural strategy and trunk muscle activation during prolonged standing in chronic low back pain patients. Gait Posture. 2015 Oct;42(4):584-9. doi: 10.1016/j.gaitpost.2015.09.008. Epub 2015 Sep 15. PMID 26404082